CLINICAL TRIAL: NCT05335460
Title: Envafolimab Combined With XELOX in Neoadjuvant Therapy for Locally Advanced Colon Cancer，A Prospective, Single Arm, Single Center ǁ Phase Clinical Trial
Brief Title: To Determine the Efficacy and Safety of Envafolimab Combined With XELOX for Locally Advanced Colon Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STEP-EX001
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Colon Cancer
Keywords: locally advanced colon cance; Envafolimab
MeSH Terms: conditions — Colonic Neoplasms | interventions — envafolimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab combined with XELOX regimen (Experimental): Envafolimab:300mg,sc,d1,Q3W XELOX( Oxaliplatin 130mg/m2,ivgtt, Q3w capecitabine 1000mg/m2, p.o Q3w)
  Interventions: Drug: Envafolimab

INTERVENTIONS:
Drug: Envafolimab — 300mg,sc,d1,Q3W
  Other Names: XELOX( Oxaliplatin 130mg/m2,ivgtt, Q3w capecitabine 1000mg/m2, p.o Q3w)

SUMMARY:
The objective is to investigate the efficacy and safety of Envafolimab combined with XELOX in neoadjuvant therapy for locally advanced colon cancer

DETAILED DESCRIPTION:
According to the 2019 NCCN guidelines, immunocheckpoint inhibitors are recommended for first-line treatment of metastatic colon cancer patients with high microsatellite instability (msi-h) or mismatched gene deletion (dMMR) who are not suitable for intensive treatment, and for all patients with second-line or above msi-h /dMMR treatment.

This study is a single-center, single-arm phase II study, patients received neoadjuvant therapy with Envafolimab combined with XELOX regimen, with one treatment cycle every 3 weeks and after two cycles accept surgery. To determine the pathologic downstage rates at time of radical resection of colon cancer following neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of colon adenocarcinoma
2. Radiological signs, evaluated by CT, of T4 or Tany N+ (AJCC 8th) 3 No metastatic involvement in other organs (M0). 4 Uncomplicated primary tumor 5 Patients who have not received systemic chemotherapy or other anti-tumor treatment 6 18-75 years； 7 ECOG 0-1； 8 The patient must have adequate organ function and meet the following laboratory test values during the screening period within 7 days before enrolling:

   * Absolute neutrophil cell count (ANC) ≥1.5x109/L, platelet ≥75x109/L, hemoglobin ≥90g/L.(in (Patients with no blood transfusion or growth factor support should be given for 7 days prior to blood collection.)
   * Serum creatinine ≤1.5× upper normal range (ULN) or estimated creatinine clearance ≥50mL/min, Glutamate aminotransferase and glutamate aminotransferase (AST and ALT)≤3×ULN.
   * Total bilirubin ≤1.5×ULN;If there is Gilbert syndrome or if the indirect bilirubin concentration indicates an extrahepatic source of bile The rise of erythrosin is ≤3×ULN.
   * Aptt ≤1.5×ULN, and INR or PT≤1.5×ULN. 9 Systemic corticosteroids or other systemic immunosuppressive drugs were used within 2 weeks prior to treatment. Immunosuppressive drugs were started or expected to be used during the trial. Inhaled corticosteroids, physiologic replacement doses of glucocorticoids are allowed 10 Sign written informed consent. 11 Expected overall survival ≥3 months 12 A person is operation and compliance with medical treatment

Exclusion Criteria:

1. Known to be allergic to any study drug
2. The patient has a history of autoimmune disease
3. Systemic corticosteroids or other systemic immunosuppressive drugs were used within 2 weeks prior to treatment.
4. The patient has severe active infections
5. A person is known to be infected with the immunodeficiency virus (HIV) or known to be HIV-positive 6、Patients Have high blood pressure that cannot be well controlled by antihypertensive medication or any other uncontrolled disease

7 pregnant women or Lactating women 8 The patient has mental illness and cannot comply with the study regulations 9 According to the judgment of the researcher, the patient have other factors that may affect the results of the study or cause the study to be terminated, such as alcohol abuse, drug abuse, other serious diseases (including mental diseases) requiring combined treatment. Patients have severe laboratory abnormalities, which will affect the safety of the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
TRG0/1 | within 7 days after surgery
  the rate of Tumor Regression Grading level 0/1

SECONDARY OUTCOMES:
R0 resection rate | within 7 days after surgery
  The tumor was completely removed, and the cutting edge was negative under microscope, without tumor residue
ORR | within 1 year after surgery
  Objective response rate

OTHER OUTCOMES:
PCR rate | within 7 days after surgery
  There were no residual tumor cells under microscope

IPD SHARING:
Plan to Share IPD: No